CLINICAL TRIAL: NCT00453206
Title: Reduced Intensity Allogeneic Hematopoietic Cell Transplantation for Patients With Hematological Diseases
Brief Title: Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer or Other Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001366; CCCWFU-29506 (Other: CCCWFU); IRB00001366 (Other: WFUHS IRB)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; blastic phase chronic myelogenous leukemia; primary myelofibrosis; chronic phase chronic myelogenous leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; de novo myelodysplastic syndromes; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; prolymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; polycythemia vera; stage III chronic lymphocytic leukemia; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent childhood anaplastic large cell lymphoma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Leukemia, Prolymphocytic; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Polycythemia Vera; Recurrence; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Extranodal NK-T-Cell | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine, busulfan, and melphalan, before a donor peripheral stem cell transplant or bone marrow transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus, methotrexate, mycophenolate mofetil, and antithymocyte globulin before and after transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer or abnormal cells as not belonging in the patient's body and destroy them (graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

PURPOSE: This phase II trial is studying how well donor stem cell transplant works in treating patients with hematologic cancer or other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility (i.e., risk of treatment-related mortality during the first 6 months after transplantation) of administering reduced-intensity allogeneic hematopoietic stem cell transplantation to patients with hematologic cancer or other diseases.

Secondary

* Determine the response rate (partial and complete response), 6- and 12-month probabilities of response, and time to progression in patients treated with this regimen.
* Determine the risk of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine other toxicities of this regimen in these patients.
* Determine the overall survival and disease-free survival of patients treated with this regimen.
* Determine the impact of iron status on overall and disease-free survival.
* Determine the influence of quality of life (at time of transplantation) on overall survival.

OUTLINE:

* Preparative regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3. Patients also receive busulfan IV over 2 hours every 6 hours on days -4 and -3 or melphalan IV over 2 hours on day -3.
* Graft-versus-host disease (GVHD) prophylaxis: Patients with matched related donors receive oral tacrolimus twice daily on days -1 to 90 followed by a taper until day 180. Patients also receive methotrexate IV on days 1, 3, and 6. Patients with matched unrelated and 9/10 matched related donors receive oral tacrolimus twice daily on days -1 to 180 followed by a taper; methotrexate IV on days 1, 3, 6, and 11; and oral mycophenolate mofetil twice daily on days -2 to 60 followed by a taper. All patients also receive antithymocyte globulin IV over 4 to 6 hours once a day on days -4 to -1.
* Allogeneic stem cell transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0. Patients receive filgrastim (G-CSF) beginning on day 7 and continuing until blood counts recover.
* Lymphocyte infusion: Patients with progressive or stable disease while off immunosuppression and no active GVHD may receive up to 3 donor lymphocyte infusions from the original donor at 8-week intervals beginning on day 180 or 210 .

Quality of life is assessed at baseline.

After completion of study therapy, patients are followed every 3 months for 2 years and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hematological disease, including any of the following:

  * Chronic lymphocytic leukemia

    * Absolute lymphocytosis > 5,000/µL
    * Morphologically mature lymphocytes with < 55% prolymphocytes
    * Lymphocyte phenotype with expression of CD19 and CD5
    * Absence of CD23 expression allowed provided disease is morphologically distinguished from mantle cell lymphoma
  * Prolymphocytic leukemia

    * Absolute lymphocytosis > 5,000/µL
    * Morphologically mature lymphocytes with > 55% prolymphocytes
  * Non-Hodgkin's or Hodgkin's lymphoma

    * Any WHO classification histologic subtype
    * Diagnosis by core biopsy allowed provided there is adequate tissue for diagnosis and immunophenotyping
    * Diagnosis by bone marrow biopsy not acceptable for follicular lymphomas
  * Multiple myeloma

    * Has received ≥ 1 prior treatment regimen
    * Has a partial response or greater by the Blade Criteria
    * Patients who achieved complete remission are eligible
  * Acute myeloid leukemia

    * Documented control (i.e., < 10% bone marrow blasts and no circulating blasts)
  * Myelodysplastic syndromes

    * Documented disease as defined by WHO or French-American-British Cooperative group criteria
    * Chronic myelogenous leukemia
  * Patients with atypical chronic myelogenous leukemia (i.e., absent Philadelphia chromosome) are eligible
  * Polycythemia vera

    * Documented disease as defined by WHO criteria (i.e., A1 + A2, and any other category A, OR A1 + A2, and any 2 category B):

      * A1: Total red blood cell mass > 25% above mean normal predicted value OR hemoglobin > 18.5 g/dL in males, 16.5 g/dL in females (hematocrit ≥ 60% in males or ≥ 56% in females)
      * A2: No cause of secondary erythrocytosis (absence of familial erythrocytosis, no elevation of epoetin alfa [EPO] due to hypoxia, high oxygen affinity hemoglobin, truncated EPO receptor, or inappropriate ectopic EPO production)
      * A3: Splenomegaly
      * A4: Clonal genetic abnormality other than the Philadelphia chromosome
      * A5: Endogenous erythroid colony formation in vitro
      * B: Platelet count > 400,000/mm³, WBC > 12,000/mm³, bone marrow biopsy with prominent erythroid and megakaryocytic proliferation, and low serum EPO
  * Chronic idiopathic myelofibrosis

    * Documented disease as defined by WHO criteria
    * Must have a HLA-identical donor, a matched unrelated donor, or a HLA 9/10 related donor meeting the following criteria:
    * HLA-identical sibling (6/6)

      * Serologic typing for class I (A, B)
      * Molecular typing for class II (DRB1)
    * 9/10 matched related donor

      * High-resolution molecular typing at HLA-A, B, C, DRB1, and DQB1
      * Only a single mismatch at one class I or II allele allowed
    * 10/10 matched unrelated donor

      * Molecular identity at HLA-A, B, C, DRB1, and DQB1 by high-resolution typing
      * Syngeneic donors are not eligible
* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* DLCO ≥ 40% with no symptomatic pulmonary disease
* LVEF ≥ 30% by cardiac MRI or echocardiogram with no symptomatic cardiac disease
* Fertile patients willing to use effective contraception

Exclusion Criteria:

* Uncontrolled diabetes mellitus
* Active serious infection
* Known hypersensitivity to E. coli-derived products
* Known HIV positivity
* History of another malignancy*, meeting the following criteria:

  * Non-skin malignancy or melanoma within the past 5 years
  * Concomitant malignancy that has not been curatively treated
  * NOTE: *However, cancer survivors who have undergone potentially curative therapy for a prior malignancy at least 5 years before enrollment and are deemed at low risk of < 30% for recurrence by their treating physicians is considered
* Pregnant or nursing

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-02; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hurd, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Intensity Allogeneic Cell Transplantation: reduced intensisty transplant are those that do not completely eliminate the patient's stem cells prior to recieving the bone marrow transplant
Period: Overall Study
Arm/Group | Reduced Intensity Allogeneic Cell Transplantation
Started | 66
Completed | 65
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Intensity Allogeneic Cell Transplantation
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality Within the First 6 Months After Transplantation
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Cell Transplantation
Number analyzed (Participants) | 65
participants | 6

2. Secondary Outcome: Complete Response
Time Frame: monthly
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Time Frame: monthly
Reporting Status: Not Posted

4. Secondary Outcome: Disease-free Survival
Time Frame: monthly
Reporting Status: Not Posted

5. Secondary Outcome: Graft-versus-host Disease
Time Frame: monthly
Reporting Status: Not Posted

6. Secondary Outcome: Iron Status at the Time of Transplantation
Time Frame: baseline
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life at the Time of Transplantation
Time Frame: baseline
Reporting Status: Not Posted

8. Secondary Outcome: Treatment-related Mortality at 100 Days After Transplantation
Time Frame: 100 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The only adverse events collected and analyzed for this study were grade 5 (death) related to transplant occurring within 6 months of transplant. No data was collected for less serious adverse events.
Arm/Group | Reduced Intensity Allogeneic Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 6/65
Other Adverse Events (participants affected / at risk) | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Allogeneic Cell Transplantation (N=65)
Graft versus host disease (Immune system disorders) | 3 (3)
Post transplant proliferative disorder (Immune system disorders) | 1 (1)
Neurological unspecified (Nervous system disorders) | 1 (1)
Death of unknown cause (General disorders) | 1 (1) — Cause of death could not be determined. Per study, this was considered related to transplant

LIMITATIONS AND CAVEATS:
By the time the primary objective of this trial was completed, the treatment approach of the trial had become standard of care. Analysis was therefore limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes